CLINICAL TRIAL: NCT04020146
Title: PPAR-γ, RXR, and VDR Expressions in Gingival Tissue Samples of Healthy Individuals, Periodontitis and Peri-implantitis Patients
Brief Title: PPAR, RXR, and VDR Expressions in Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, mehmet murat taskan, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: Gaziosmanpasa University
Record Dates: First submitted 2019-07-08; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis; Periimplantitis
Keywords: periodontitis; periimplantitis; RXR; VDR
MeSH Terms: conditions — Periodontitis; Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1;: healthy controls (C, n=15),
  Interventions: Other: Gingival biopsies
- group 2: periodontitis patients with stage 3 grade B; (P, n=15)
  Interventions: Other: Gingival biopsies
- group 3: peri-implantitis patients (PI, n=15).
  Interventions: Other: Gingival biopsies

INTERVENTIONS:
Other: Gingival biopsies — Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processing.

SUMMARY:
ABSTRACT Objective: Periodontitis and peri-implantitis are the irreversible destructive diseases of the periodontal and peri-implant tissues. The present study aimed to determine the receptor expressions of Peroxisome proliferative-activated receptor (PPAR)-γ, Retinoid X receptor (RXR)-α, and Vitamin D receptor (VDR) in the diseased tissues around teeth and dental implants.

Methods: The study consisted of three groups as group 1; healthy controls (C, n=15), group 2; periodontitis patients with stage 3 grade B (P, n=15), and group 3; peri-implantitis patients (PI, n=15). Periodontal clinical parameters as the plaque index (PI), gingival index (GI) and clinical attachment levels (CAL) were recorded. Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processing. Hematoxylin-eosin (H&E) and immunohistochemistry staining were performed. Total inflammatory cell counts and fibroblast cell density were evaluated on H&E-stained slides while PPAR-γ, RXR-α, and VDR were evaluated via immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* periodontitis patients
* periimplantitis patients

Exclusion Criteria:

* smokers,
* systemically compromised patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study consisted of three groups as group 1; healthy controls (C, n=15), group 2; periodontitis patients with stage 3 grade B (P, n=15), and group 3; peri-implantitis patients (PI, n=15).
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory cells counts | 6 months
  Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processing. Hematoxylin-eosin (H&E) staining were performed. Total inflammatory cell counts density were evaluated on H&E-stained slides.A cell counting frame of 10.000 µm2 area was selected under 1000x magnification. The total inflammatory cells (neutrophil, lymphocyte, eosinophil, and macrophage cells) within the frame were counted as inflammatory cell counting.
Fibroblast counts | 6 months
  Fibroblasts counts were evaluated from H&E stained slides under 1000x magnification via a light microscope (Nikon Eclipse, E 600, Tokyo, Japan).
Peroxisome proliferative-activated receptor (PPAR)-γ | During histological processing
  Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processin and immunohistochemistry staining were performed, PPAR-γ, was evaluated via immunohistochemistry. Samples were examined under 400x magnification using light microscopy (Nikon Eclipse, E 600, Tokyo, Japan).
Retinoid X receptor (RXR)-α | 6 months
  Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processing and immunohistochemistry staining were performed, RXR-α was evaluated via immunohistochemistry. Samples were examined under 400x magnification using light microscopy (Nikon Eclipse, E 600, Tokyo, Japan).
Vitamin D receptor (VDR) | 6 months
  . Gingival biopsies were obtained from all participants and biopsy samples underwent histological tissue processing and immunohistochemistry staining were performed, VDR was evaluated via immunohistochemistry. Samples were examined under 400x magnification using light microscopy (Nikon Eclipse, E 600, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No